CLINICAL TRIAL: NCT03622528
Title: Precision, Pulmonary Disease Evaluation and Lung Cancer Detection Using Quantitative Low-dose CT
Brief Title: Quantitative Lung Cancer Screening
Status: Withdrawn | Type: Observational
Why Stopped: Funding Issues
Sponsor: Jessica Sieren (Other)
Collaborators: Vida Diagnostics, Inc (Unknown)
Responsible Party: Sponsor-Investigator, Jessica Sieren, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201603824
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Pulmonary Disease; Chronic Obstructive Pulmonary Disease; Cancer, Lung
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Lung Cancer Screening Cohort: Patients who are seen in the UIHC lung cancer screening clinic will be asked to undergo an additional standard chest CT scan during their UIHC clinical lung cancer screening CT scan. Additionally, data from that clinical scan and all medical records associated with nodules that were discovered by the Lung Cancer Screening, will also be collected.
  Interventions: Radiation: Chest CT scan

INTERVENTIONS:
Radiation: Chest CT scan — Standard dose chest CT scan

SUMMARY:
The purpose of this project is to validate quantitative lung structure assessment using an automated analysis software (VIDA), for application to low dose computed tomography (LDCT) acquired for lung cancer screening. Currently the software runs on standard dose CT data. In addition, it is the plan to incorporate algorithms into the software to address assessment of any identified pulmonary lesions.

DETAILED DESCRIPTION:
The purpose of this project is to validate quantitative lung structure assessment using an automated analysis software (VIDA), for application to low dose computed tomography (LDCT) acquired for lung cancer screening. Currently the software runs on standard dose CT data. In addition, it is the plan to incorporate algorithms into the software to address assessment of any identified pulmonary lesions.

The Lung Cancer Screening Clinic is a new program that screens a group of patients that meet a predetermined criteria, set by the program, for lung cancer. At this time primary care providers, within the UIowa network, have the ability to place an order for this screening process for their patients. The hope is to expand this program to any primary care provider in the future. Clinic staff look over the patients past medical history to determine if they fit the clinic criteria.

For this study, the study team will ask the patients seen in the lung cancer screening clinic at the University of Iowa to undergo an additional standard dose CT scan during that same visit(for comparison/validation of the software performance). For those subjects that agree to participate, the study team will also ask to collect the data and CT scans that were also collected for their clinical Lung Cancer Screening visit. For this group the study team will also ask to collect all medical records associated with nodules found at this Lung Cancer Screening visit.

The study team propose to test the performance of VIDA's existing image analysis tools for the assessment of chronic obstructive pulmonary disease (COPD), when applied to the LDCT data acquired for lung cancer screening. The study team will also develop new lung nodule evaluation functions to specifically address the clinical needs within the at-risk lung cancer patient population.

To carry out the work, the study team propose two specific aims:

1. Validate VIDA's quantitative computed tomography (QCT) metrics for COPD and emphysema utilizing the lung cancer LDCT screening cohort as compared to the standard quantitative high resolution computed tomography (HRCT) scanning protocol. With collaboration between the University of Iowa and VIDA, the study team will establish a tightly controlled, CT data acquisition protocol in our local lung cancer screening program. Data collected will incorporate thin-slice and iterative reconstructions, breath coaching to target lung inflation levels for patients and HRCT data acquisition in a sub-cohort. The VIDA analysis will be refined and the appropriate reconstruction setting identified such that the outputs from the LDCT data correlate to the HRCT (current standard) outputs.
2. Complete and refine development of VIDA's novel lung nodule segmentation algorithm for solid and non-solid nodules using the standardized lung cancer LDCT screening protocol. Automated nodule segmentation in CT scans is challenging due to border ambiguity with neighboring structures (such as vessels and the pleura), poor boundary contrast of more subtle nodules, and noise associated with LDCT. The study team will develop a novel method that robustly segments pulmonary lesions by allowing mutual interaction between the nodules and surrounding structures, leading to a highly accurate segmentation with less manual corrective actions for a high volume lung cancer screening workflow.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that meet the clinical Lung Cancer Screening guidelines and participate in that clinical screening.

Exclusion Criteria:

* Subjects that do not meet the clinical Lung Cancer Screening guidelines.

Ages: 50 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects will be patients at the University of Iowa Hospitals and Clinics that are participating in the Lung Cancer Screening clinic and have met those guidelines for being included in that screening program.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Segmental Airway Branch Differences | 1 day of Study Visit
  Segmental airway branch differences will be measured by comparing the clinical low dose chest CT scan and the standard dose chest CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sieren, PhD, Principal Investigator — University of Iowa